CLINICAL TRIAL: NCT06699407
Title: Efficacy and Safety of Qishenyiqi Dripping Pills in Patients With Ventricular Remodeling and Chronic Heart Failure With Reduced Ejection Fraction After Myocardial Infarction
Brief Title: Qishenyiqi for Ventricular Remodeling After Myocardial Infarction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Qishenyiqi and HFrEF
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Chronic Stable Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qishenyiqi (Experimental)
  Interventions: Drug: Qishenyiqi dripping pills
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qishenyiqi dripping pills — Qishenyiqi dripping pills, 1 bag once, three times a day, 12 months
  Arms: Qishenyiqi
Drug: Placebo — Placebo, 1 bag once, three times a day, 12 months
  Arms: Placebo

SUMMARY:
The effects of Qishenyiqi dripping pill on cardiac remodeling in patients with chronic stable heart failure have not been reported. This project aims to clarify the efficacy and safety of Qishenyiqi in patients with chronic heart failure after myocardial infarction. Patients with chronic stable heart failure after myocardial infarction were selected and randomly divided into two groups: the treatment group was treated with Qishenyiqi dripping pills; The control group was given placebo treatment. After 12 months of follow-up, the effects of Qishenyiqi on cardiac remodeling and function and cardiovascular adverse events were evaluated. The results are helpful to provide a new treatment strategy for chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* 1) The history of acute myocardial infarction exceeds 3 months;
* 2) Symptoms and signs of heart failure have been stable for more than one month;
* 3) 18 years old or more;
* 4) NYHA cardiac function classified as grade II~IV;
* 5) LVEF≤40%；
* 6) NT-proBNP≥450pg/ml；
* 7) All subjects or their guardians must sign the subject consent before entering the trial.

Exclusion Criteria:

* 1) Patients with the following diseases: nonischemic cardiomyopathy; valvular heart disease; congenital heart disease; obstruction of left ventricular outflow tract; severe decompensated heart failure; active myocarditis or pericardial disease; end-stage liver and kidney diseases; malignant tumor;
* 2) Planned to undergo cardiac surgery within 12 months;
* 3) Mechanical complications of myocardial infarction;
* 4) Pregnant or nursing, or having the intention to give birth within one year;
* 5) Patients who participated in clinical research of other drugs within 3 months before being selected;
* 6) Patients with poor sound transmission windows are examined by transthoracic ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
LVEDVI=LVEDV/BSA | From baseline to 12 months after follow-up
  Changes of left ventricular end-diastolic volume index (LVEDVI) compared with baseline after 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Panpan Hao, Jinan, Shandong
  - Qianfoshan Hospital, Shandong University, Jinan, Shandong
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan

IPD SHARING:
Plan to Share IPD: Undecided